CLINICAL TRIAL: NCT03052751
Title: A Multicenter, Randomized, Investigator- and Subject-Blind, Placebo-Controlled, Treatment Sequence Study Evaluating the Safety, Tolerability, and Efficacy of UCB7665 in Subjects With Moderate to Severe Myasthenia Gravis
Brief Title: Study to Test the Safety, Tolerability and Efficacy of UCB7665 in Subjects With Moderate to Severe Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG0002; 2016-002698-36 (EudraCT Number)
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Myasthenia Gravis
Keywords: UCB7665; Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — rozanolixizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is an Investigator- and Subject-Blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dosage Regimen 1 (Experimental): Subjects randomized in dosage regimen 1 will receive 3 doses of UCB7655 (dose 1) in dosing period 1 and will then be re-randomized into dosing period 2 to receive 3 doses of UCB7665 (dose 1 or dose 2).
  Interventions: Drug: UCB7665
- Dosage Regimen 2 (Experimental): Subjects randomized in dosage regimen 2 will receive 3 doses of placebo in dosing period 1 and will then be re-randomized into dosing period 2 to receive 3 doses of UCB7665 (dose 1 or dose 2).
  Interventions: Drug: UCB7665; Other: Placebo

INTERVENTIONS:
Drug: UCB7665 — UCB7665 will be administered in 2 different dosages (dose 1 and dose 2). UCB7665 (INN: Rozanolixizumab) is a humanized monoclonal antibody that is being developed for treatment of IgG autoantibody-mediated conditions such as myasthenia gravis (MG)
  Other Names: Rozanolixizumab
Other: Placebo — Placebo will be administered in period 1 of dosage regimen 2.
  Arms: Dosage Regimen 2

SUMMARY:
The purpose of the study is to evaluate the clinical efficacy of UCB7665 as a chronic-intermittent treatment in subjects with generalized myasthenia gravis (MG) who are classified as moderate to severe.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a well-documented diagnosis of myasthenia gravis (MG) at Visit 1 (Screening), based on subject history and supported by previous evaluations
* Subject would currently be considered for treatment with immunological therapy (immunoglobulin/plasma exchange (IVIG/PLEX)) by the investigator
* Subject has a well-documented record of autoantibodies against anti-acetylcholine receptor (Anti-AChR) or anti-muscle specific kinase (Anti-MuSK) prior to Screening
* Female subjects must either be: postmenopausal, permanently sterilized or if childbearing potential applicable will use a highly effective method of birth control
* Male subjects must be willing to use a method of contraception

Exclusion Criteria:

* Subject has previously received treatment in this study or subject has previously been exposed to UCB7665
* Subject has participated in another study of an investigational medicinal product (IMP; or a medical device) within the previous 30 days of Screening or is currently participating in another study of an investigational medicinal product (IMP; or a medical device)
* Subject has a known hypersensitivity to any components of the IMP
* Subject has a history of hyperprolinemia, since L-proline is a constituent of the UCB7665 IMP
* Subjects with Myasthenia Gravis (MG) only affecting the ocular muscles
* Subjects with severe weakness affecting oropharyngeal or respiratory muscles, or who have myasthenic crisis at Screening or impending crisis
* Subject has quantitative myasthenia gravis (QMG) score of <11 at Baseline
* Subject has a serum total immunoglobulin G (IgG) level <= 6g/L at Screening
* Absolute neutrophil count <1500 cells/mm^3
* Subject has any medical condition (acute or chronic illness) or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the subject's ability to participate in this study
* Subject has any laboratory abnormality that, in the opinion of the investigator, is clinically significant, has not resolved at randomization, and could jeopardize or would compromise the subject's ability to participate in this study
* Subject has received a live vaccination within 8 weeks prior to the Baseline Visit; or intends to have a live vaccination during the course of the study or within 7 weeks following the final dose of IMP
* Subject has received any experimental biological agent within or outside of a clinical study in the past 3 months or within 5 half-lives prior to Baseline (whichever is longer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 877 822 9493 (UCB)
Locations (20):
- United States (6):
  - Mg0002 712, Los Angeles, California
  - Mg0002 701, Orange, California
  - Mg0002 713, Miami, Florida
  - Mg0002 708, Tampa, Florida
  - Mg0002 707, Augusta, Georgia
  - Mg0002 704, Columbus, Ohio
- Belgium (3):
  - Mg0002 102, Brussels
  - Mg0002 103, Ghent
  - Mg0002 101, Leuven
- Canada (3):
  - Mg0002 203, London
  - Mg0002 202, Montreal
  - Mg0002 201, Toronto
- Mg0002 302, Ostrava-Poruba, Czechia
- Denmark (2):
  - Mg0002 401, Aarhus
  - Mg0002 402, Copenhagen
- Germany (3):
  - Mg0002 505, Düsseldorf
  - Mg0002 502, Gummersbach
  - Mg0002 501, Jena
- Spain (2):
  - Mg0002 601, Barcelona
  - Mg0002 602, Barcelona

REFERENCES:
- [Derived] Matic A, Alfaidi N, Bril V. An evaluation of rozanolixizumab-noli for the treatment of anti-AChR and anti-MuSK antibody-positive generalized myasthenia gravis. Expert Opin Biol Ther. 2023 Jul-Dec;23(12):1163-1171. doi: 10.1080/14712598.2023.2296126. Epub 2023 Dec 28. PMID 38099334
- [Derived] Regnault A, Morel T, de la Loge C, Mazerolle F, Kaminski HJ, Habib AA. Measuring Overall Severity of Myasthenia Gravis (MG): Evidence for the Added Value of the MG Symptoms PRO. Neurol Ther. 2023 Oct;12(5):1573-1590. doi: 10.1007/s40120-023-00464-x. Epub 2023 May 11. PMID 37166675
- [Derived] Bril V, Benatar M, Andersen H, Vissing J, Brock M, Greve B, Kiessling P, Woltering F, Griffin L, Van den Bergh P; MG0002 Investigators. Efficacy and Safety of Rozanolixizumab in Moderate to Severe Generalized Myasthenia Gravis: A Phase 2 Randomized Control Trial. Neurology. 2021 Feb 9;96(6):e853-e865. doi: 10.1212/WNL.0000000000011108. Epub 2020 Nov 20. PMID 33219142
- [Derived] Smith B, Kiessling A, Lledo-Garcia R, Dixon KL, Christodoulou L, Catley MC, Atherfold P, D'Hooghe LE, Finney H, Greenslade K, Hailu H, Kevorkian L, Lightwood D, Meier C, Munro R, Qureshi O, Sarkar K, Shaw SP, Tewari R, Turner A, Tyson K, West S, Shaw S, Brennan FR. Generation and characterization of a high affinity anti-human FcRn antibody, rozanolixizumab, and the effects of different molecular formats on the reduction of plasma IgG concentration. MAbs. 2018 Oct;10(7):1111-1130. doi: 10.1080/19420862.2018.1505464. Epub 2018 Sep 12. PMID 30130439

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in May 2017 and concluded in August 2018.
Pre-assignment Details: The Participant Flow refers to the Randomized Set (RS) which consisted of all participants randomized into the study at the first randomization visit.
Groups:
- Placebo: Participants received 3 doses of placebo in Dosing Period 1 and then were re-randomized into Dosing Period 2 to receive 3 doses of UCB7665 (7 mg/kg or 4 mg/kg).
- UCB7665 (7 mg/kg): Participants received 3 doses of UCB7665 (7 mg/kg) in Dosing Period 1 and then were re-randomized into Dosing Period 2 to receive 3 doses of UCB7665 (7 mg/kg or 4 mg/kg).
- Placebo - UCB7665 (7 mg/kg): Participants randomized to receive 3 doses of placebo at weekly intervals in Dosing Period 1 were then re-randomized to receive 3 doses of UCB7665 (7 mg/kg) at weekly intervals in Dosing Period 2.
- Placebo - UCB7665 (4 mg/kg): Participants randomized to receive 3 doses of placebo at weekly intervals in Dosing Period 1 were then re-randomized to receive 3 doses of UCB7665 (4 mg/kg) at weekly intervals in Dosing Period 2.
- UCB7665 (7 mg/kg) - UCB7665 (7 mg/kg): Participants randomized to receive 3 doses of UCB7665 (7 mg/kg) at weekly intervals in Dosing Period 1 were then re-randomized to receive 3 doses of UCB7665 (7 mg/kg) at weekly intervals in Dosing Period 2.
- UCB7665 (7 mg/kg) - UCB7665 (4 mg/kg): Participants randomized to receive 3 doses of UCB7665 (7 mg/kg) at weekly intervals in Dosing Period 1 were then re-randomized to receive 3 doses of UCB7665 (4 mg/kg) at weekly intervals in Dosing Period 2.
Period: Dosing Period 1
Arm/Group | Placebo | UCB7665 (7 mg/kg) | Placebo - UCB7665 (7 mg/kg) | Placebo - UCB7665 (4 mg/kg) | UCB7665 (7 mg/kg) - UCB7665 (7 mg/kg) | UCB7665 (7 mg/kg) - UCB7665 (4 mg/kg)
Started | 22 | 21 | 0 | 0 | 0 | 0
Completed Period 1 | 22 | 21 | 0 | 0 | 0 | 0
Completed Period 1 and Started Period 2 | 22 | 20 | 0 | 0 | 0 | 0
Completed | 22 | 20 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Period: Dosing Period 2
Arm/Group | Placebo | UCB7665 (7 mg/kg) | Placebo - UCB7665 (7 mg/kg) | Placebo - UCB7665 (4 mg/kg) | UCB7665 (7 mg/kg) - UCB7665 (7 mg/kg) | UCB7665 (7 mg/kg) - UCB7665 (4 mg/kg)
Started | 0 | 0 | 11 | 11 | 10 | 10
Completed | 0 | 0 | 8 | 11 | 10 | 10
Not Completed | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 0 | 0 | 0
Period: Observation Period
Arm/Group | Placebo | UCB7665 (7 mg/kg) | Placebo - UCB7665 (7 mg/kg) | Placebo - UCB7665 (4 mg/kg) | UCB7665 (7 mg/kg) - UCB7665 (7 mg/kg) | UCB7665 (7 mg/kg) - UCB7665 (4 mg/kg)
Started | 22 | 21 | 11 | 11 | 10 | 10
Completed | 22 | 21 | 11 | 11 | 9 | 10
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set (RS) which consisted of all participants randomized into the study at the first randomization visit.
Arm/Group | Placebo | UCB7665 (7 mg/kg) | Total Title
Number analyzed (Participants) | 22 | 21 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 18 | 32
  >=65 years | 8 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (15.7) | 50.5 (14.7) | 51.9 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black | 1 | 1 | 2
  White | 19 | 20 | 39
  Other/mixed | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Quantitative Myasthenia Gravis (QMG) Score to Visit 9
Description: The total QMG score was obtained by summing the responses to each individual item (13 items; Responses: None=0, Mild=1, Moderate=2, Severe=3). The score ranges from 0 to 39, with lower scores indicating lower disease activity. The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Visit 9 (up to Day 29)
Population: The FAS consisted of all participants in the SS who had a Baseline and at least 1 post-Baseline QMG measurement during Dosing Period 1 (up to and including Visit 9, ie, Day 29).
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Placebo (FAS): Participants received 3 doses of placebo in Dosing Period 1. Participants formed the Full Analysis Set (FAS) which consisted of all participants in the Safety Set (SS) who had a Baseline and at least 1 post-Baseline QMG measurement during Dosing Period 1 (up to and including Visit 9, ie, Day 29).
- UCB7665 (7 mg/kg) (FAS): Participants received 3 doses of UCB7665 (7 mg/kg) in Dosing Period 1. Participants formed the Full Analysis Set (FAS) which consisted of all participants in the Safety Set (SS) who had a Baseline and at least 1 post-Baseline QMG measurement during Dosing Period 1 (up to and including Visit 9, ie, Day 29).
Arm/Group | Placebo (FAS) | UCB7665 (7 mg/kg) (FAS)
Number analyzed (Participants) | 22 | 21
scores on a scale | -1.2 (0.6) | -1.8 (0.6)
Statistical Analysis 1: Comparison: Placebo (FAS) vs UCB7665 (7 mg/kg) (FAS); Mixed Model Repeated Measures (MMRM) Analysis of Covariance (ANCOVA) model included fixed terms for treatment group, visit, interaction between treatment group and visit, covariate of Baseline QMG score, and random effect for participant. The differences presented was 'UCB7665 (7 mg/kg) minus Placebo'; Test type: Superiority; p = 0.221, MMRM — One-sided p-value was presented for difference; LS Mean Difference vs Placebo = -0.7, 95% CI 1-sided [upper limit 0.8] — Estimate included treatment and treatment by visit interaction effects

2. Secondary Outcome: Change From Baseline in Myasthenia Gravis-Composite Score to Visit 9
Description: The total Myasthenia Gravis (MG)-composite score was obtained by summing the responses to each individual item (10 items; Grade: 0-9 depending on item). The score ranges from 0 to 50, with lower scores indicating lower disease activity. The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Visit 9 (up to Day 29)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | UCB7665 (7 mg/kg) (FAS)
Number analyzed (Participants) | 22 | 21
scores on a scale | -1.2 (0.9) | -3.1 (0.9)
Statistical Analysis 1: Comparison: Placebo (FAS) vs UCB7665 (7 mg/kg) (FAS); MMRM ANCOVA model included fixed terms for treatment group, visit, interaction between treatment group and visit, covariate of Baseline MG-composite score, and random effect for participant. The differences presented was 'UCB7665 (7 mg/kg) minus Placebo'; Test type: Superiority; p = 0.089, MMRM — One-sided p-value was presented for difference; LS Mean Difference vs Placebo = -1.8, 95% CI 1-sided [upper limit 0.4] — Estimate included treatment and treatment by visit interaction effects

3. Secondary Outcome: Change From Baseline in Myasthenia Gravis-Activities of Daily Living (MGADL) Score to Visit 9
Description: The total MGDAL score was obtained by summing the responses to each individual item (8 items; Grades: 0, 1, 2, 3). The score ranges from 0 to 24, with lower scores indicating lower disease activity. The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Visit 9 (up to Day 29)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | UCB7665 (7 mg/kg) (FAS)
Number analyzed (Participants) | 22 | 21
scores on a scale | -0.4 (0.5) | -1.8 (0.5)
Statistical Analysis 1: Comparison: Placebo (FAS) vs UCB7665 (7 mg/kg) (FAS); ANCOVA model included fixed terms for treatment group, covariate of Baseline MGADL score; Test type: Superiority; p = 0.036, ANCOVA — One-sided p-value was presented for difference; LS Mean Difference vs Placebo = -1.4, 95% CI 1-sided [upper limit -0.1] — Estimate included treatment effect

ADVERSE EVENTS:
Time Frame: From the start of Treatment Period at Baseline and up to Observation Period at 8 weeks after the final dose of IMP.
Groups:
- Placebo (SS): Participants received 3 doses of placebo in Dosing Period 1 and then were re-randomized into Dosing Period 2 to receive 3 doses of UCB7665 (7 mg/kg or 4 mg/kg). Participants formed the Safety Set (SS) which consisted of all participants in the Randomized Set (RS) who had received at least 1 dose of investigational product (IMP).
- UCB7665 (7 mg/kg) (SS): Participants received 3 doses of UCB7665 (7 mg/kg) in Dosing Period 1 and then were re-randomized into Dosing Period 2 to receive 3 doses of UCB7665 (7 mg/kg or 4 mg/kg). Participants formed the Safety Set (SS) which consisted of all participants in the Randomized Set (RS) who had received at least 1 dose of investigational product (IMP).
- Placebo - UCB7665 (7 mg/kg) (SS): Participants randomized to receive 3 doses of placebo at weekly intervals in Dosing Period 1 were then re-randomized to receive 3 doses of UCB7665 (7 mg/kg) at weekly intervals in Dosing Period 2. Participants formed the Safety Set (SS).
- Placebo - UCB7665 (4 mg/kg) (SS): Participants randomized to receive 3 doses of placebo at weekly intervals in Dosing Period 1 were then re-randomized to receive 3 doses of UCB7665 (4 mg/kg) at weekly intervals in Dosing Period 2. Participants formed the Safety Set (SS).
- UCB7665 (7 mg/kg) - UCB7665 (7 mg/kg) (SS): Participants randomized to receive 3 doses of UCB7665 (7 mg/kg) at weekly intervals in Dosing Period 1 were then re-randomized to receive 3 doses of UCB7665 (7 mg/kg) at weekly intervals in Dosing Period 2. Participants formed the Safety Set (SS).
- UCB7665 (7 mg/kg) - UCB7665 (4 mg/kg) (SS): Participants randomized to receive 3 doses of UCB7665 (7 mg/kg) at weekly intervals in Dosing Period 1 were then re-randomized to receive 3 doses of UCB7665 (4 mg/kg) at weekly intervals in Dosing Period 2. Participants formed the Safety Set (SS).
Arm/Group | Placebo (SS) | UCB7665 (7 mg/kg) (SS) | Placebo - UCB7665 (7 mg/kg) (SS) | Placebo - UCB7665 (4 mg/kg) (SS) | UCB7665 (7 mg/kg) - UCB7665 (7 mg/kg) (SS) | UCB7665 (7 mg/kg) - UCB7665 (4 mg/kg) (SS)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21 | 0/11 | 0/11 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/22 | 0/21 | 3/11 | 1/11 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 7/22 | 13/21 | 7/11 | 9/11 | 8/10 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=22) | UCB7665 (7 mg/kg) (SS) (N=21) | Placebo - UCB7665 (7 mg/kg) (SS) (N=11) | Placebo - UCB7665 (4 mg/kg) (SS) (N=11) | UCB7665 (7 mg/kg) - UCB7665 (7 mg/kg) (SS) (N=10) | UCB7665 (7 mg/kg) - UCB7665 (4 mg/kg) (SS) (N=10)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myasthenia gravis crisis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=22) | UCB7665 (7 mg/kg) (SS) (N=21) | Placebo - UCB7665 (7 mg/kg) (SS) (N=11) | Placebo - UCB7665 (4 mg/kg) (SS) (N=11) | UCB7665 (7 mg/kg) - UCB7665 (7 mg/kg) (SS) (N=10) | UCB7665 (7 mg/kg) - UCB7665 (4 mg/kg) (SS) (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Infusion site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammatory pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (5) | 12 (22) | 3 (4) | 2 (2) | 4 (5) | 4 (6)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Myasthenic syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT03052751/Prot_002.pdf
  • Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT03052751/SAP_003.pdf